CLINICAL TRIAL: NCT06963437
Title: Comparison of Revisional Surgery, Ketogenic Diet, and Intermittent Fasting in Bariatric Surgery Patients With Weight Regain: A Prospective Randomized Controlled Study
Brief Title: Interventions for Weight Regain After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Seher Dallı Şen, Seher Dallı Şen, PhD Candidate in Nutrition and Dietetic, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEDU-SBE-SS-01
Record Dates: First submitted 2025-04-18; First posted 2025-05-09 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Obese Patients With Bariatric Surgery; Obese Patients (BMI ≥ 30 kg/m²); Weight Regain Post Bariatric Surgery; Revisional Bariatric Surgery; Ketogenic Dieting; Intermittent Fasting
Keywords: weight regain post bariatric surgery; revisional bariatric surgery; ketogenic dieting; intermittent fasting; nutritional status
MeSH Terms: conditions — Intermittent Fasting | interventions — Diet; Diet, Ketogenic; Angptl4 protein, mouse; Control Groups

STUDY DESIGN:
Intervention Model Description: This study will be conducted on 56 patients who have experienced insufficient weight loss (IWL) or weight regain (WR) following bariatric surgery. Participants will be randomly assigned to one of four groups (n=14 per group):
  RBS Group - patients undergoing revisional bariatric surgery (RBS)
  VLCKD Group - patients following a very low-calorie ketogenic diet (VLCKD)
  IF Group - patients following an intermittent fasting (IF) diet
  Control Group - patients receiving standard post-bariatric nutritional follow-up as recommended by the ASMBS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Revisional bariatric surgery (RBS) group (Experimental): A nutrition program in accordance with ASMBS guidelines will be implemented for patients undergoing revisional bariatric surgery.
  Interventions: Other: Diet
- Very low-calorie ketogenic diet (VLCKD) group (Experimental): The daily energy intake of VLCKD will be planned as 600-800 kcal, with approximately 10% of energy from carbohydrates (<30 g/day), 40-45% from protein, and 40-50% from fat.
  Interventions: Other: Ketogenic diet
- Intermittent fasting (IF) group (Experimental): Time-restricted intermittent fasting (16/8) will be applied. Patients in this group will follow a feeding schedule limited to an 8-hour window (16/8) for a duration of 6 weeks.
  Interventions: Other: Fasting
- Control group (Active Comparator): No individualized diet will be planned; instead, patients will receive education on the stage 4 dietary guidelines recommended for lifelong adherence following bariatric surgery.
  Interventions: Other: Control

INTERVENTIONS:
Other: Diet — A four-stage dietary program will be implemented in accordance with ASMBS guidelines. To the best of our knowledge, there is currently no study comparing the dietary approach following revisional bariatric surgery with ketogenic and intermittent fasting diets
  Other Names: bariatric diet
  Arms: Revisional bariatric surgery (RBS) group
Other: Ketogenic diet — A high-protein Very Low-Calorie Ketogenic Diet (VLCKD) will be implemented as the nutritional intervention. In line with previous studies, the daily energy intake of the ketogenic diet will be planned as 600-800 kcal, with approximately 10% of energy from carbohydrates (<30 g/day), 40-45% from protein, and 40-50% from fat. Total carbohydrate intake will be restricted to less than 30 g per day, primarily from vegetables, while fat intake will derive from natural protein sources and 10 g of olive oil per day.
  Arms: Very low-calorie ketogenic diet (VLCKD) group
Other: Fasting — Patients in this group will follow a time-restricted eating pattern (16/8) for a duration of 6 weeks, with food intake limited to an 8-hour window each day. Intermittent fasting will preferably be observed between 6:00 PM and 10:00 AM; however, patients may choose alternative 16-hour fasting periods such as 7:00 PM-11:00 AM or 8:00 PM-12:00 PM, depending on their individual routines. During the 8-hour feeding window, patients will adhere to the stage 4 post-bariatric dietary guidelines in accordance with ASMBS recommendations
  Other Names: intermittent fasting
  Arms: Intermittent fasting (IF) group
Other: Control — No individualized diet will be planned
  Other Names: Control Group
  Arms: Control group

SUMMARY:
Study Objective:

The aim of this study is to evaluate the effects of revisional bariatric surgery (RBS), very low-calorie ketogenic diet (VLCKD), and intermittent fasting (IF) on nutritional habits and clinical outcomes (anthropometric and biochemical measurements) in patients with insufficient weight loss (IWL) or weight regain (WR) after bariatric surgery, and to compare these findings with those of a control group.

DETAILED DESCRIPTION:
Study Hypotheses:

1. In patients with IWL or WR after bariatric surgery, a diet following the bariatric care guidelines (BCGs) after revisional bariatric surgery (RBS) improves nutritional habits, anthropometric, and biochemical parameters.
2. In patients with IWL or WR after bariatric surgery, VLCKD improves nutritional habits, anthropometric, and biochemical parameters.
3. In patients with IWL or WR after bariatric surgery, IF regimen improves nutritional habits, anthropometric, and biochemical parameters.
4. In patients with IWL or WR after bariatric surgery, the diet program recommended by the ASMBS as part of standard post-bariatric care improves nutritional habits, anthropometric measurements, and biochemical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 45 years who have undergone bariatric surgery (BS).
* Experiencing inadequate weight loss (IWL) within 18 months after surgery or weight regain (WR) following successful weight loss.
* Definitions used in the study:

IWL is defined as <50% excess weight loss (EWL) 18 months postoperatively. WR is defined as >25% regain of the lost weight (from the lowest achieved weight).

-

Exclusion Criteria:

* Pregnant or lactating women.
* Patients with acute illnesses, infections, or comorbidities that may affect treatment efficacy or safety (e.g., cancer, type 1 diabetes, renal or hepatic failure, recent stroke or myocardial infarction, nephrolithiasis, substance or alcohol abuse, eating disorders, severe depression or other psychiatric disorders, inflammatory bowel disease, neoplasms, arrhythmic heart diseases, heart failure, respiratory failure).
* Patients currently receiving corticosteroid therapy.
* Professional athletes.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight (kg) | Baseline and Week 6
  Body weight will be measured at baseline and at Week 6 using a calibrated digital scale while participants are wearing light clothing and no shoes. Statistical analyses will be performed using SPSS v22.0. Normality will be tested using Shapiro-Wilk. ANOVA or Kruskal-Wallis will be used as appropriate; p<0.05 considered significant.
Change in Body Mass Index (kg/m²) | Baseline and Week 6
  BMI will be calculated as weight (kg) divided by the square of height (m²), using body weight and height measurements obtained with a digital scale and a wall-mounted stadiometer.
  Statistical analyses will be performed using SPSS v22.0. Normality will be tested using Shapiro-Wilk. ANOVA or Kruskal-Wallis will be used as appropriate; p<0.05 considered significant.
Change in Waist Circumference (cm) | Baseline and Week 6
  Waist circumference will be measured using a non-elastic measuring tape while participants are standing upright. The measurement will be taken 5 cm below the umbilicus.
  Statistical analyses will be performed using SPSS v22.0. Normality will be tested using Shapiro-Wilk. ANOVA or Kruskal-Wallis will be used as appropriate; p<0.05 considered significant.
Change in Body Composition (Fat Mass %, Muscle Mass %,) assessed by BIA | Baseline and Week 6
  Body composition parameters, including fat mass (%), fat-free mass (%), muscle mass (%), and ECW/TBW ratio, will be assessed using multi-frequency segmental bioelectrical impedance analysis (BIA) (Tanita MC-780 MA, Korea). Assessments will follow ESPEN guidelines.
  Statistical analyses will be performed using SPSS v22.0. Normality will be tested using Shapiro-Wilk. ANOVA or Kruskal-Wallis will be used as appropriate; p<0.05 considered significant.
Percentage Weight Loss (%WL) | Baseline and Week 6
  %WL will be calculated using the formula: [(Preoperative weight - Postoperative weight) / Preoperative weight] × 100
Percentage Excess Weight Loss (%EWL) | Baseline and Week 6
  %EWL will be calculated using the formula: [(Preoperative weight - Postoperative weight) / (Preoperative weight - Ideal weight)] ×100 *Ideal weight is defined as the weight corresponding to a BMI of 25 kg/m².*

SECONDARY OUTCOMES:
Change in Fasting Blood Glucose (mg/dL) | Baseline and Week 6
  Fasting venous blood samples will be collected after an overnight fast of at least 8 hours, both at baseline and at Week 6. Fasting blood glucose will be measured using standardized automated analyzers in a certified clinical laboratory.
  Descriptive statistics will be reported as mean ± SD or median (min-max). Group comparisons will be made using ANOVA or Kruskal-Wallis, with significance set at p<0.05.
Change in Fasting Insulin (µIU/mL) | Baseline and Week 6
  Serum insulin concentrations will be determined from fasting blood samples taken at baseline and Week 6 using standardized laboratory methods.
  Descriptive statistics will be reported as mean ± SD or median (min-max). Group comparisons will be made using ANOVA or Kruskal-Wallis, with significance set at p<0.05.
Change in Lipid Profile (HDL, LDL, Total Cholesterol, Triglycerides) (mg/dL) | Baseline and Week 6
  Lipid levels will be assessed from fasting blood samples. The lipid profile includes high- density lipoprotein (HDL), low-density lipoprotein (LDL), total cholesterol, and triglycerides.
  Descriptive statistics will be reported as mean ± SD or median (min-max). Group comparisons will be made using ANOVA or Kruskal-Wallis, with significance set at p<0.05.
Change in Renal Function Markers (BUN, Creatinine, Uric Acid, Urea) (mg/dL) | Baseline and Week 6
  Renal function parameters will be analyzed using fasting blood samples to determine changes in blood urea nitrogen (BUN), creatinine, uric acid, and urea levels.
  Descriptive statistics will be reported as mean ± SD or median (min-max). Group comparisons will be made using ANOVA or Kruskal-Wallis, with significance set at p<0.05.
Change in Liver Function Tests (ALT, AST, Albumin, Total Protein) (U/L, g/dL) | Baseline and Week 6
  Liver function will be assessed by measuring serum levels of alanine aminotransferase (ALT), aspartate aminotransferase (AST), albumin, and total protein.
  Descriptive statistics will be reported as mean ± SD or median (min-max). Group comparisons will be made using ANOVA or Kruskal-Wallis, with significance set at p<0.05.
Change in Vitamin and Mineral Status (Vitamin B12, Folic Acid, Magnesium, Calcium, Sodium, Potassium) (ng/L, mg/dL, mmol/L, etc.) | Baseline and Week 6
  Serum concentrations of vitamins and minerals will be measured from fasting samples. Parameters include vitamin B12, folic acid, magnesium, total calcium, sodium, and potassium.
  Descriptive statistics will be reported as mean ± SD or median (min-max). Group comparisons will be made using ANOVA or Kruskal-Wallis, with significance set at p<0.05.
Change in Hematological Parameters (Hemoglobin, Hematocrit, Ferritin, Serum Iron, TIBC) (g/dL, µg/L, etc.) | Baseline and Week 6
  Hematological status will be evaluated using fasting blood samples to assess hemoglobin, hematocrit, ferritin, serum iron, and total iron binding capacity (TIBC).Descriptive statistics will be reported as mean ± SD or median (min-max). Group comparisons will be made using ANOVA or Kruskal-Wallis, with significance set at p<0.05.
Change in Daily Energy and Macronutrient Intake | Baseline and Week 6
  Daily intake of energy (kcal/day) and macronutrients-protein, fat, carbohydrate, and fiber (g/day)-will be assessed using 3-day dietary records (including one weekend day) and a validated Food Frequency Questionnaire (FFQ). Data will be analyzed using BEBIS-9 (Nutrition Information System, Turkey). Dietary records will be reviewed for completeness and accuracy by trained dietitians. Results will be reported in kcal/day and g/day.
  Descriptive statistics will be reported as mean ± SD or median (min-max). Group comparisons will be made using ANOVA or Kruskal-Wallis, with significance set at p<0.05.
Change in Micronutrient Intake | Baseline and Week 6
  Micronutrient intake (e.g., vitamins and minerals) will be assessed using 3-day dietary records and the FFQ. Data will be analyzed using BEBIS-9, with results reported in standard units (e.g., mg/day, µg/day). Intake values will be interpreted in relation to dietary reference values but without applying a composite scoring scale.
  Descriptive statistics will be reported as mean ± SD or median (min-max). Group comparisons will be made using ANOVA or Kruskal-Wallis, with significance set at p<0.05.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Özel Nev FSM Hastanesi, Bursa, Bursa
  - Özel Nev FSM Hastanesi, Nilufer, Bursa

IPD SHARING:
Plan to Share IPD: No
Due to ethical and privacy considerations, individual participant data will not be shared